CLINICAL TRIAL: NCT07354633
Title: Full Sail Ahead, Sailing in Psychosocial Rehabilitation.
Acronym: VOILE_RPS93
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Raluca ROSETTI, MBBS, psychiatrist and investigator, Centre hospitalier de Ville-Evrard, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VOILE_RPS93_10477M
Record Dates: First submitted 2025-11-28; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Disorder
Keywords: Sailing; psychiatric disorder; physical conditions
MeSH Terms: conditions — Mental Disorders | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: one group is voile and the other one is control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sailing arm (Active Comparator): 20 users followed in the psychosocial rehabilitation unit (UNIRRE 93) and practicing the sailing activity by session of 10 sailing sessions over two periods (March to June and August to November) Twice a year (month)
  Interventions: Behavioral: sailing
- control (Placebo Comparator): 20 control subjects: users followed in the psychosocial rehabilitation unit (UNIRRE 93) and taken care of in psychosocial rehabilitation without a veil over the same period as a "veil" session.
  Interventions: Behavioral: taking care in rehabilitation psychosocial

INTERVENTIONS:
Behavioral: sailing — Users followed in the psychosocial rehabilitation unit (UNIRRE 93) and practicing the sailing activity by session of 10 sailing sessions over two periods (March to June and August to November) Twice a year (month)
  Arms: sailing arm
Behavioral: taking care in rehabilitation psychosocial — control subjects: users followed in the psychosocial rehabilitation unit (UNIRRE 93) and taken care of in psychosocial rehabilitation without a veil over the same period as a "veil" session.
  Arms: control

SUMMARY:
This study is part of the desire to develop disabled sports in the territory of Seine-Saint-Denis and responds to the national strategy plan Sport Santé, 2019-2024, which addresses all audiences. The law of January 26, 2016 recognizes sport as a non-drug therapeutic in its own right, becoming an element of the hospital care pathway but also ambulatory. The partnership between the EPS of Ville-Evrard and the departmental committee of Voile du 93, co-funder of the project thus allows the diversification and the increase of the offer of care in psychosocial rehabilitation.

DETAILED DESCRIPTION:
Sailing is integrated into the psychosocial rehabilitation offer for people with severe psychological disorders, for example in Italy . Since 2021, the Psychosocial Rehabilitation Reference Unit (UNIRRE 93) of the Ville-Evrard hospital has been using sailing as a therapeutic intervention. After 4 years of implementation within the psychosocial rehabilitation referral unit in Seine-Saint-Denis, this innovative care needs to be evaluated and shared within the psychiatric care community. This study is part of the desire to develop disabled sports in the territory of Seine-Saint-Denis and responds to the national strategy plan Sport Santé, 2019-2024, which addresses all audiences.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining free and informed consent to the research project
* User over 18 years old and living in the 93
* Living with a psychic or neurodevelopmental disorder
* Supported by the RPS 93 platform
* Have obtained a medical certificate of fitness for sailing including competition (only for the sailing group)
* Knowing French language ( how to read and write)
* Clinical condition stabilized for less than three months despite taking medication

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Psychiatric decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
scale of quality of life | T0: before sailing starts
  The questionnaire is a validated health-related quality of life scale. The scale is also recommended by the HAS to evaluate clinical practices. It is composed of 36 elements, including eight scales focusing on health: general physical state, limitations of roles related to physical health, body pain, general perception of health, vitality, social functioning, limitations of roles related to mental health. The scale can be auto or hetero administered and requires 5 to 10 minutes of handover.
Scale of quality of life | T1: within 10 minutes after the end of sailing
  The questionnaire is a validated health-related quality of life scale. The scale is also recommended by the HAS to evaluate clinical practices. It is composed of 36 elements, including eight scales focusing on health: general physical state, limitations of roles related to physical health, body pain, general perception of health, vitality, social functioning, limitations of roles related to mental health. The scale can be auto or hetero administered and requires 5 to 10 minutes of handover.
Scale of quality of life | T2: Three months After Sailing
  The questionnaire is a validated health-related quality of life scale. The scale is also recommended by the HAS to evaluate clinical practices. It is composed of 36 elements, including eight scales focusing on health: general physical state, limitations of roles related to physical health, body pain, general perception of health, vitality, social functioning, limitations of roles related to mental health. The scale can be auto or hetero administered and requires 5 to 10 minutes of handover.
Warwick Edinburgh mental well being scale | T0: Before sailing starts
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated tool designed to measure mental wellbeing in individuals and populations, consisting of 14 positively worded items scored on a 5-point Likert scale.All items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item answered on a 1 (Never) to 5 (All the time) Likert scale. The minimum scale score is 14 and the maximum is 70. Higher scores indicate better mental well being.
Warwick Edinburgh mental well being scale | T1: within 10 minutes after the end of sailing
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated tool designed to measure mental wellbeing in individuals and populations, consisting of 14 positively worded items scored on a 5-point Likert scale.All items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item answered on a 1 (Never) to 5 (All the time) Likert scale. The minimum scale score is 14 and the maximum is 70. Higher scores indicate better mental well being.
Warwick Edinburgh mental well being scale | T2: Three months After Sailing
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated tool designed to measure mental wellbeing in individuals and populations, consisting of 14 positively worded items scored on a 5-point Likert scale.All items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item answered on a 1 (Never) to 5 (All the time) Likert scale. The minimum scale score is 14 and the maximum is 70. Higher scores indicate better mental well being.
Self-Esteem Scale | T0: before sailing starts
  Rosenberg's Self-esteem Scale By Nathalie Crépin and Florence Delerue Self-esteem is defined as the judgment or evaluation one makes of oneself, of one's value personal. In a simpler way, self-esteem can also be assimilated to self-affirmation. Esteem of oneself is an essential factor in sports performance.This scale represents a French cross-cultural validation of the Rosenberg Self-Esteem Scale (1965). It contains 10 items, five positive and five negative assessed on a 1 to 4-point scale It takes only 8 minutes to do the scale.
Self-Esteem Scale | T1: within 10 minutes after the end of sailing
  Rosenberg's Self-esteem Scale By Nathalie Crépin and Florence Delerue Self-esteem is defined as the judgment or evaluation one makes of oneself, of one's value personal. In a simpler way, self-esteem can also be assimilated to self-affirmation. Esteem of oneself is an essential factor in sports performance.This scale represents a French cross-cultural validation of the Rosenberg Self-Esteem Scale (1965). It contains 10 items, five positive and five negative assessed on a 1 to 4-point scale It takes only 8 minutes to do the scale.
Self-Esteem Scale | T2: Three months After Sailing
  Rosenberg's Self-esteem Scale By Nathalie Crépin and Florence Delerue Self-esteem is defined as the judgment or evaluation one makes of oneself, of one's value personal. In a simpler way, self-esteem can also be assimilated to self-affirmation. Esteem of oneself is an essential factor in sports performance.This scale represents a French cross-cultural validation of the Rosenberg Self-Esteem Scale (1965). It contains 10 items, five positive and five negative assessed on a 1 to 4-point scale It takes only 8 minutes to do the scale.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Rusheenthira Thavaseelan, Neuilly-sur-Marne
  - EPS VIlle Evrard - UNIRRE 93, Neuilly-sur-Marne

IPD SHARING:
Plan to Share IPD: No